CLINICAL TRIAL: NCT06839638
Title: Efficacy of Trichloroacetic Acid (100%) Versus Cryotherapy in Patients with Xanthelasma Palpebrarum
Brief Title: Efficacy of 100% Trichloroacetic Acid Vs. Cryotherapy in Xanthelasma Palpebrarum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Amra Batool, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NishtarMU2
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Xanthelasma Palpebrarum
Keywords: Hyperlipidemia-related Skin Lesions; Non-Surgical Treatment for Xanthelasma; Chemical Cauterization
MeSH Terms: conditions — Xanthomatosis | interventions — Trichloroacetic Acid; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group TCA (Experimental): will receive 100% TCA application to xanthelasma lesions using the dipstick method.
  Interventions: Procedure: 100% Trichloroacetic Acid (TCA)
- Group Cryotherapy (Active Comparator): will receive cryotherapy using liquid nitrogen. A single freeze-thaw cycle will be performed until a narrow halo of white ice forms around the lesion.
  Interventions: Procedure: Cryotherapy (Liquid Nitrogen)

INTERVENTIONS:
Procedure: 100% Trichloroacetic Acid (TCA) — Patients in this group will receive 100% TCA application to xanthelasma lesions using the dipstick method. The surrounding skin will be protected with white soft paraffin to prevent chemical spillage. Post-treatment, Fusidic acid 2% will be applied twice daily for one week. Treatment efficacy will be assessed after six weeks.
  Arms: Group TCA
Procedure: Cryotherapy (Liquid Nitrogen) — Patients in this group will receive cryotherapy using liquid nitrogen. A single freeze-thaw cycle will be performed until a narrow halo of white ice forms around the lesion. Post-treatment care will include Fusidic acid 2% applied twice daily for one week. Treatment efficacy will be assessed after six weeks.
  Arms: Group Cryotherapy

SUMMARY:
Xanthelasma palpebrarum (XP) is a common skin condition characterized by yellowish plaques that typically develop around the eyelids. While not harmful, these plaques can be a cosmetic concern for many individuals. Several treatment options exist, but there is no clear consensus on the most effective method.

This study aims to compare the effectiveness of two treatment options-100% trichloroacetic acid (TCA) and cryotherapy-in removing xanthelasma palpebrarum. Trichloroacetic acid is a chemical solution that removes the lesions by controlled cauterization, while cryotherapy involves freezing the plaques using liquid nitrogen.

A total of 60 patients with xanthelasma will be randomly assigned to receive either 100% TCA or cryotherapy. The success of the treatment will be determined based on whether the plaques flatten and disappear within six weeks. The results of this study will help identify the more effective treatment method, which can be used to improve patient outcomes and minimize recurrence.

The study is being conducted at Nishtar Hospital Multan and aims to provide valuable insights for dermatologists in choosing the best treatment for xanthelasma palpebrarum.

DETAILED DESCRIPTION:
Xanthelasma palpebrarum (XP) is a common dermatological condition characterized by the presence of yellowish plaques around the inner canthus of the eyelids. While benign, these plaques are often a significant cosmetic concern for patients. Various treatment modalities are available, including surgical excision, laser therapy, electrocauterization, chemical cauterization with trichloroacetic acid (TCA), and cryotherapy. However, each treatment option has its limitations, including variable efficacy, risk of recurrence, and potential side effects. Despite the availability of multiple therapeutic approaches, no consensus exists regarding the most effective and cosmetically acceptable treatment for XP.

This randomized controlled trial aims to compare the efficacy of 100% trichloroacetic acid (TCA) versus cryotherapy (liquid nitrogen) for the treatment of xanthelasma palpebrarum. TCA is a commonly used chemical cauterizing agent that causes epidermal necrosis, leading to the sloughing of lipid-laden histiocytes responsible for XP formation. Cryotherapy, on the other hand, involves the application of extreme cold to induce tissue destruction, promoting lesion resolution. Both modalities are non-surgical, cost-effective, and relatively simple to perform, making them viable options for outpatient dermatological treatment.

Sixty patients with xanthelasma palpebrarum will be enrolled in the study and randomly allocated into two treatment groups. Group A will receive 100% TCA application using the dipstick method, ensuring controlled application while protecting the surrounding skin with white soft paraffin. Group B will be treated with cryotherapy, using a single freeze-thaw cycle with liquid nitrogen until a narrow halo of white ice forms around the lesion. Following the procedure, all patients will apply Fusidic acid 2% twice daily for one week as post-treatment care.

The primary outcome measure will be the complete resolution of xanthelasma, assessed at six weeks after treatment through clinical examination and photographic documentation. The study will also evaluate secondary outcomes, including post-treatment adverse effects such as hypopigmentation, erythema, ulceration, and scarring. A blinded consultant dermatologist will assess treatment response and determine efficacy based on predefined criteria.

This study is particularly significant as there is currently no published comparative study from South Punjab evaluating these two treatment modalities. By providing evidence on the relative efficacy and safety of TCA and cryotherapy, this research will help dermatologists select the most effective, safe, and cosmetically acceptable treatment for XP. The findings may also contribute to future treatment guidelines, improving patient outcomes and reducing the need for retreatment in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-55 years
* Either male or female
* No prior treatment for xanthelasma palpebrarum (XP)
* Patients on anti-lipidemic drugs for systemic control of disease
* Bilateral xanthelasmas measuring between 0.5 cm to 3 cm

Exclusion Criteria:

• History of hypersensitivity to TCA or cryotherapy.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 100% Trichloroacetic Acid (TCA) versus Cryotherapy in Xanthelasma Palpebrarum | Six weeks after treatment initiation
  Complete disappearance and flattening of xanthelasma plaques, assessed through clinical examination by a blinded dermatologist.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, Principal Investigator — Nishtar Hospital, Multan
Locations (1):
- Nishtar Hospital, Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No